CLINICAL TRIAL: NCT05910346
Title: The Effect of Training and Counseling Based on Mercer's Maternal Role Theory on Maternal Attachment and Maternal Function: A Randomized Controlled Study
Brief Title: The Effect of Training and Counseling Based on Mercer Maternal Role Theory on Maternal Attachment and Maternal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: KAMİLE ALTUNTUĞ (Unknown)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, Lecturer, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mercer
Record Dates: First submitted 2023-06-04; First posted 2023-06-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Maternal-Fetal Relations; Maternal Behavior
Keywords: maternal identity, maternal role, being a mother
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In order to prevent statistical bias, data analysis will be performed by an independent statistician, and the experimental and control groups specified as A and B during the analysis will not be shared with the statistician. Intention-to-treat analysis-ITT will be performed at the end of the study in order to prevent the reduction bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): At the beginning of the study, the pregnant women who applied to the obstetrics clinics and met the sample selection criteria will be divided into the experimental and control groups by randomization method by filling out the Personal Information Form. Motherhood Theory-Based Education Program will be applied to the pregnant women who are allocated to the experimental group.
  Interventions: Behavioral: education and counseling based on maternal role theory
- Control Group (No Intervention): First stage: Pregnant women in the control group will receive routine care. Second stage: Data Collection Form for the follow-up and Birth Process and Results will be filled within the first 24 hours after the birth.
  Third stage: Follow-up will be done by phone within 4 weeks after birth. Maternal Attachment Scale (MBI), Barkin Maternal Function Inventory will be applied.
  Fourth stage: At the end of the fourth month postpartum, follow-up counseling will be made by telephone and the Maternal Attachment Scale and the Barkin Maternal Function scale will be filled.
  Fifth stage: When the study is completed, a training booklet will be given to the mothers in the control group.

INTERVENTIONS:
Behavioral: education and counseling based on maternal role theory — Pregnant women in the experimental group will be given training and counseling based on the maternal role theory, starting at 32 weeks of gestation (1 week in total, 2 days a week, 3 sessions every day, 6 sessions in total, 8 hours in total). After the training and counseling program given to the pregnant women in the experimental group according to the motherhood role theory is completed, a training booklet will be prepared so that they can repeat the information they have learned until birth (for improving the motherhood role). It is planned to give the training booklet at the end of the training in order to ensure continuity in the program.
  Arms: Experimental Group

SUMMARY:
Motherhood role gain is the composition of social roles and developmental behaviors and attitudes that continue with the formation of motherhood identity development in the postnatal period that started during pregnancy. In many studies, it is stated that mothers should be prepared to transition to motherhood roles in the prenatal period in order to enable them to develop successful motherhood identity. This study will be carried out to determine the effect of structured birth preparation education on the material attachment status and motherhood function according to the theory of motherhood. The study was planned as a single -blind, post -test parallel group randomized controlled experimental study. The universe of the study will form pregnant women who apply to Necmettin Erbakan University Meram Medical Faculty Hospital Birth and Gynecology Polyclinic and Clinic. When the sample of the study was calculated as 95 %confidence interval, 5 %error and 80 %power, a total of 44 cases, 22 for the experimental group and 22 for the control group were found to be suitable for statistical analyzes. In this study, assuming that the loss rates in the literature will be 20 %loss when reference, 28 to the experimental group and 28 to the control group will be included in the initially 56 pregnant studies. The data will be collected using the 'Personal Information Form, Postpartum Period Features Information Form, Maternal Binding Scale and Barkin Maternity Function Inventory. Pregnant women in the experimental group will start in the 32nd gestational week and will be given structured training and counseling according to the theory of motherhood. Pregnant women in the control group will take standard care. Number, percentage, average and standard deviation analysis will be used for descriptive statistics. Parametric and nonparametric tests will be applied according to the compliance of the data for the normal distribution of the data in the study pattern in independent groups and recurrent tests. The results will be tested at P <0.05 significance level. In order to collect the data, Ethical Permission was obtained by the Decision No. 2022/024 from the Ethics Committee of KTO Karatay University Pharmaceutical and Medical Research. Necmettin Erbakan University Meram Medical Faculty Hospital will be obtained from the institution. Before starting to work, verbal and written permissions will be obtained by reading the voluntary information form to all pregnant women. Maternal attachment inventory and Barkin Motherhood Function Scale Writers were permitted via e-mail.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate,
* Between the ages of 18-35,
* At the 30nd week of pregnancy and above,
* Having a single and healthy fetus,
* Pregnant women who are open to communication and cooperation

Exclusion Criteria:

* Having a risky pregnancy history (pregnancies under 18 and over 35 years of age, EDT, PROM, Preeclampsia, Eclampsia, Epilepsy, GDM)
* Having a treatment pregnancy (mothers who became pregnant with ART),
* Having a chronic disease (DM, HT, Asthma, Epilepsy, Autoimmune diseases, self-report),
* Having a psychiatric illness (based on self-report and clinical diagnosis),
* Foreign nationals,
* Living outside the province of Konya,
* Pregnant women who participated in any childbirth preparation training program

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 56 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Maternal attachment | 1-4 mounth
  Maternal attachment will be assessed with the Maternal Attachment Inventory. As the score obtained from the scale increases, attachment increases.
Maternal function | 1-4 mounth
  Maternal function will be assessed with the Barkin Maternal Functioning Inventory. As the score obtained from the scale increases, attachment increases.attachment scale. As the score obtained from the scale increases, attachment increases.ores of educational practice based on maternal role theory during pregnancy may change.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No